CLINICAL TRIAL: NCT01388400
Title: Enriched Environments for Stroke Rehabilitation; Pilot Study to Determine Appropriate Outcome Measures and Their Sensitivity to Different Training Protocols
Brief Title: Enriched Environments for Upper Limb Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Ministry of Health, Israel (Other Government)
Responsible Party: Dr. Harold Weingarden, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-08-5120-HW-CTIL
Record Dates: First submitted 2011-06-12; First posted 2011-07-06 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; virtual reality; upper limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional intervention for upper limb reaching (Experimental): Reaching or holding cones, cups, etc. in all planes with and without gravity or loading
  Interventions: Other: conventional occupational therapy
- VR treatment (Experimental): The Virtual Reality (VR) therapy group received the treatment in the GestureTek VR environment which focused on reaching movements of the affected upper limb using virtual games and a virtual supermarket.
  Interventions: Device: video capture virtual reality

INTERVENTIONS:
Other: conventional occupational therapy — upper limb exercises
  Arms: Conventional intervention for upper limb reaching
Device: video capture virtual reality — virtual reality delivered uppe limb exercises
  Arms: VR treatment

SUMMARY:
Stroke contributes significantly to the incidence of disabilities, with upper limb (UL) motor impairment being especially prevalent. Animal studies suggest that post-stroke motor recovery is largely attributable to adaptive plasticity in brain motor areas. While some environmental training factors contributing to plastic mechanisms have been identified in animals, translation of this knowledge to the clinical setting is insufficient. Optimal recovery may be related to both external (e.g., feedback type) and internal factors (e.g., cognitive ability, motivation). Clinically feasible methods for training are needed. Use of enriched virtual environments (VEs) may provide a way to address these needs. Outcome measures that best reflect recovery need to be identified since this is an essential step to evaluate the effect of novel training programs for UL motor recovery in stroke.

The research question is which clinical and kinematic outcome measures best reflect motor performance recovery after a targeted upper limb treatment intervention. Aim 1 is to compare changes in outcome measures recorded before and after an upper limb intervention in stroke subjects to motor performance in healthy subjects. Aim 2 is to determine motor performance between-group differences sample size is based on knowledge of expected outcome measure mean score differences between groups. Hypothesis. 1: Specific clinical and kinematic outcome measures will be sensitive to within-group (pre-post intervention training) changes. Hypothesis. 2: Specific clinical and kinematic outcome measures will be sensitive to between-group (healthy vs. patients in enriched vs. conventional intervention groups. Sixteen chronic stroke survivors and 8 age- and sex-matched healthy controls will participate. Patients will be matched on cognitive and motor impairment levels and divided into two groups. Using an single subject (A-B-A) research design, kinematics during two pre-tests, 3 weeks apart, will be recorded for test-retest reliability. Stroke groups will practice varied upper limb reaching movements (15 45-minute sessions in 3 weeks) in environments providing different motivation/feedback levels. Pre- and post motor performance evaluations will be done with clinical tests and a Test Task with specific motor performance requirements. A Transfer Task will also be recorded. By comparing data analysis methods (3-Dimensional (3D) analysis of different markers or placements), the investigators will identify which kinematic outcome measures best reflect motor improvement in post-test and follow-up sessions (retention).

The expected results are identification of two primary and two secondary outcome measures that reflect upper limb motor recovery and can distinguish between motor recovery and compensation. The results will be used to design a randomized control trial to determine the efficacy of VE-based treatment on arm motor recovery. The goal is to determine how extrinsic (environmental) and intrinsic (personal) motivational factors affect motor learning in stroke survivors with cognitive and physical impairment. Knowledge gained can also be used for rehabilitation of other neurological and orthopedic pathologies.

DETAILED DESCRIPTION:
A. Scientific Background

Stroke is the third leading cause of death in Western countries and upper limb (UL) sensorimotor dysfunction contributes significantly to the incidence of physical disabilities and handicaps (Olsen 1990). One explanation for poor arm recovery is the focus on task accomplishment rather than performance quality. This may reinforce alterative (compensatory) movement strategies instead of encouraging the reappearance of pre-morbid movement patterns (recovery). Although the rehabilitative goal is recovery of function, whether this is achieved through true motor recovery or compensation is still under debate. Indeed, for some patients with severe impairment, compensation should be encouraged to maximize functional ability. Alternatively, for those with good prognosis, motor recovery is emphasized for several reasons. First, given appropriate training, recovery can continue well into the chronic stage of stroke (e.g., Michaelsen & Levin 2004). Second, while compensation may assist immediate performance, it may lead to longer-term problems such as pain and contracture (Ada et al. 1994; Levin 1997). Third, permitting compensations could encourage learned nonuse limiting the capacity for subsequent motor gains (Allred et al. 2005). While performance gains have been documented after repetitive training of isolated movements (e.g., Whitall et al. 2000), few studies have addressed whether patients can use explicit information to optimize motor skill acquisition and whether true behavioural recovery occurs. Points to consider in developing optimal training programs is that learning occurs when participants are motivated, practice a variety of related tasks and are given relevant feedback (Nudo & Friel 1999; Winstein et al. 1999). In addition, patients may not benefit from variable practice until missing motor elements are recovered (Carr & Shepherd 1987) and motor relearning is related to physical and cognitive impairment level (Cirstea et al. 2006).

To date, most studies have used only clinical measures to evaluate functional change (e.g., Jang et al. 2003) without considering how movement is performed. This study will focus on the ability to distinguish between whether functional improvement results from an increase in compensation or from true motor recovery. This can only be done by correlating functional improvement (clinical measures) with changes in arm motor patterns through detailed movement analysis (kinematics). Since there are a large number of possible kinematic indicators of improvement, the investigators need to identify which measures are most indicative of change. This is a first step in the determination of clinically meaningful outcome measures to be used in randomized control trials of the effectiveness of interventions. Clinical salience is essential to translate knowledge from research studies to evidence-based practice (van Peppen et al. 2007).

B. Study Design: 1. Detailed Plan of the Study

Two groups of 8 stroke subjects will participate in an A-B-A design in which data from post-intervention (within one week of the completion of the intervention) and follow-up (one month after the completion of the intervention)tests will be compared to data from two pre-tests (held at beginning and end of the first week of the study just prior to the start of the intervention). Multiple clinical and kinematic motor performance outcomes will be measured to determine which ones best describe arm motor recovery. This will be done by comparing changes in outcomes before and after training to mean scores of 8 age- and gender-matched healthy volunteers (recorded in a single session). Stroke survivors will practice movement in two different training environments providing different levels of motivation and feedback: Training Environment 1 will be created in a 2D video-based VR environment that will provide high motivation, Knowledge of Results (KR) about motor outcome (i.e., speed, precision) and non-specific Knowledge of Performance (KP) feedback about trunk movement. Environment 2 will be created in a physical environment that provides only KP feedback but no KR or additional motivation.

Training Protocol: After baseline evaluations (physical & cognitive), stroke groups will practice pointing to 6 standardized targets placed just beyond reach (12 trials per target) during an acquisition phase of 15 sessions spaced over three weeks (3 sessions/wk, 72 trials/session). This practice regimen incorporates elements necessary for optimal motor learning: 1) Varied practice: Although the movements are not new motor tasks, they should be re-acquired during stroke recovery. Our aim is not teach subjects a novel task but to identify how a movement performed sub-optimally may be improved with practice. 2) Intensive practice: The number of repetitions per session was chosen according to studies by Cirstea and Levin (2000). Thus, 72 trials per session (3 blocks of 24 trials, 5 min rest between blocks) are considered as 'intensive' practice, which is a necessary element for a successful training program. Following the acquisition phase, evaluations which will be repeated after 3mos to evaluate retention and transfer of motor skills.

2. Methods: Subjects Eight stroke subjects per group will be recruited. They will be matched for age and for initial arm motor severity (± 5 pts on the Fugl-Meyer Arm Assessment). Eight age- and sex-matched healthy subjects will be recruited as a control group.

Subject Recruitment: Patients will be recruited from Haim Sheba Hospital discharge lists using a procedure in place since 2005. Screening will be done by clinical research associates. Potential participants meeting inclusion criteria 1-3 and exclusion criteria will be sent an explanatory letter inviting them to contact study investigators. Informed consent will be obtained from each participant. Control subjects will be recruited from the community.

Training Environments: Motivation and Feedback: Training will be done in the Dept. of Occupational Therapy located at the Sheba Medical Center. Training environments will allow us to evaluate the effect of combining different degrees of motivation and feedback on motor outcome. Environment 1 is highly motivating (novel and fun) since training is presented as a game in which the learner tries to beat his own score in subsequent sessions. Targets are presented as balls in a video-based VR system (Gesture Xtreme). The patient sits in front of a 36 inch display of the 6 target scene. The patient's image is captured by a video camera and inserted into the scene displayed on the monitor. The task is to point to each of the targets which appear in a random sequence. Feedback will provide pertinent information for motor learning (KR, KP, game score). Environment 2 incorporates the same number and disposition of targets as Env. 1 but they will be presented in a physical environment on a wooden frame in front of the subject. KR and KP feedback will be provided as verbal cues by the experimenter as is done usually in the clinic. However, they will be no additional motivational information (game score).

Preliminary Outcome Measures: Clinical Before and after training in both stroke groups, blinded evaluators will measure clinical scores of arm motor impairment and function (Fugl-Meyer Arm Score, Reaching Performance Scale, Box and Blocks test, Wolf Motor Function Test, Motor Activity Log) as well as cognitive function. All tests are valid and reliable and are regularly used in clinical practice.

Kinematic testing: Test Task and Transfer Task:

The investigators will also record kinematic outcome measures characterizing arm and trunk movements during reaching (elbow extension, shoulder horizontal adduction, shoulder flexion, scapular movements, trunk displacement).

Our aim is to focus on segmental and joint kinematics during a Test and a Transfer Task consisting of reaching movements. Test Task will be recorded. The Test target will be placed in line with the patient's sternum at a distance just beyond the subject's arm length. The Test Task is similar to movements made to one of the practiced targets. To assess motor learning, the investigators will determine if elements learned in one task transfer to other similar tasks. Thus, the investigators will also assess movements made in a Transfer Task, to a target placed in front of the ipsilateral shoulder 5 centimeters (cm) higher than the topmost row of trained targets. The Transfer Task is therefore a new movement, not practiced during the training. Rigid body segmental kinematics will be recorded from sets of 4 passive reflective markers (0.5 cm diameter spheres) attached to the trunk, upper arm and forearm segments. This will enable the computation of three translational and three rotational degrees of freedom per segment. Joint kinematics will be collected from markers fixed on the sternum, acromion, elbow and wrist via exo-skeletal frames. Marker motion will be recorded with a calibrated 3 camera opto-electronic motion-capture system (ProReflex MCU-240, Qualisys) on suitable computer software (Qualisys, Göteborg, Swe). Data collection (100 Hertz, 2-5 seconds) will be triggered by movement of the hand from a central position by release of a mechanical switch. The accuracy of the measurements of each marker is within an error of <0.2 cm.

As a first step, the investigators will determine movement times, accuracy, smoothness, segment and joint rotations and the main components of multi-joint coordination. Cartesian coordinates (x,y,z) for each segment will be obtained from the segmental marker sets. Raw data from at least three markers per segment will be used after interpolation of missing markers (5th-order polynomial). For each trial, movement times and peak velocities will be determined from endpoint tangential velocity traces. Movement time is the time between the point at which the tangential velocity exceeds and remains above 5% of its maximum and then returns to and remains below this level. Movement accuracy in terms of constant extent errors will be computed as the mean distance (d) between the final endpoint position (x, y, z) and the position of the target (x0, y0, z0). Constant and variable (SD) directional errors will also be defined. Movement smoothness will be computed from the tangential velocity trace using the index of curvature (ratio of endpoint path length to length of a straight line joining the initial and final positions) and the number of peaks in the trajectory path. For segment and joint rotations, vectors will be calculated within reference coordinate systems for the upper and forearm segments.

From the resulting segment centroid motion and segment rotation data different outcome variables will be calculated. The most relevant ones will define changes in performance with respect to the endpoint motion and with respect to the whole-arm posture, particularly, the evolution of the movement over time (time derivatives) and the fragmentation of the segmental path and posture of the arm while moving towards the different targets. Additional aspects of movement will be explored in order to find the most appropriate descriptors of arm motor performance and changes after the proposed clinical interventions.

Change scores will be calculated for each subject to determine an Index of Improvement (IP) and an Index of Learning (IL). The IP is defined as the change in each variable as a ratio of post- to pre-test values. An IP of 1 indicates no change whereas negative and positive values indicate that the value decreased or increased respectively. For some variables, positive ratios will indicate improvement (endpoint velocity, endpoint smoothness, angle measures, phase amplitudes) while for others, improvement will be demonstrated by negative ratios (movement time, movement precision). The IL, used to determine if subjects retain improvements after training for each follow-up epoch, is defined as the change in the variable at retention- compared to post-test. IL values of 1 indicate that the improvement is maintained (no change), of negative value that the parameter decreased and of positive value that the parameter increased.

Statistical analysis: For our first aim, changes in outcome measures will be determined by comparing movement outcomes before and after the acquisition and retention phases by two-repeated measures mixed design ANOVA (MANOVA) and comparing raw means (Time 1, Time 2, Time 3, Time 4) and change scores (IP, IL) between groups. The investigators will determine which kinematic measures undergo the most change and thus may be most indicative of motor recovery (e.g., increase in elbow and/or shoulder movement, decrease in trunk movement) by investigating which measures are the most different between training groups. The investigators expect changes in the group training in Environment I to be greater than those in from the group training in Environment 2.

ELIGIBILITY:
Inclusion Criteria for patients wth stroke:

1. Age 40-80 years
2. sustained a single stroke between 3-24 months prio t study leading to upper limb paresis
3. have at least Stage 3/7 arm control (mild to moderate motor deficits) on the Chedoke-McMaster Scale.
4. <81 yrs old to minimize confounding effects of age-related changes in sensorimotor functions

Exclusion Criteria for patients wth stroke:

1. other neurological or orthopaedic problems that may interfere with interpretation of results
2. significant deficits in attention, constructional skills, neglect and apraxia
3. shoulder subluxation, arm pain
4. lack of endurance as judged by a physician
5. undergoing other therapy, surgery or medical procedures within the study period.

Inclusion Criteria for healthy control subjects:

1. Age 40-80 years

Exclusion Criteria for control subjects:

1. any neurological or orthopaedic problems that may interfere with interpretation of results.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Post test Wolf Motor Function Test | Change from baseline after 3 week treatment intervention
  Wolf Motor Function Test (WMFT; Wolf et al., 1989) assessed upper limb motor function (quality and speed) on 15 functional tasks scored on 6-point (0-5) scales as well as 2 strength (grip strength and resistance while lifting or moving weighted objects) measures (Wolf et al., 2001). The tasks are arranged in order of increasing complexity and progress from proximal to distal joint involvement. The WMFT has high interrater (Interclass Correlation Coefficient =0.97-0.99), as well as test-retest reliability (0.90 for performance time and 0.95 for performance quality).
Follow-up Wolf Motor Function Test | Change from baseline 4 weeks after end of treatment intervention
  Wolf Motor Function Test (WMFT; Wolf et al., 1989) assessed upper limb motor function (quality and speed) on 15 functional tasks scored on 6-point (0-5) scales as well as 2 strength (grip strength and resistance while lifting or moving weighted objects) measures (Wolf et al., 2001). The tasks are arranged in order of increasing complexity and progress from proximal to distal joint involvement. The WMFT has high interrater (Interclass Correlation Coefficient =0.97-0.99), as well as test-retest reliability (0.90 for performance time and 0.95 for performance quality).

SECONDARY OUTCOMES:
Post test Fugl-Meyer Arm Scale | Change from baseline after 3 week treatment intervention
  Fugl-Meyer Arm Scale (FMA; Fugl-Meyer, 1975) was developed to assess active motor function after stroke, based on the stages of recovery described by Twitchell and Brunnstrom (Sanford et al., 1993). Movements are scored between 0-2 points, and the summary score ranges from 0 (complete paralysis) to 66 (full ROM). The assessment has high validity (Berglund and Fugl-Meyer 1986) and reliability (Duncan et al. 1983) composite test-retest = 0.98-0.99; Interclass Correlation Coefficient for interrater reliability=0.96, p<0.0001; internal reliability = 90.7%) (Wolf et al., 2001).
Post test Composite Spasticity Index | Change from baseline after 3 week treatment intervention
  Composite Spasticity Index (CSI, Levin and Hui-Chan, 1992) assessed phasic (tendon jerk, clonus) and tonic (resistance to stretch) reflex responses in the elbow flexors when the limb was stretched at a moderate speed (>100/second). The valid (Nadeau et al. 1997) and reliable (Goulet et al. 1996) composite score ranges from 0 to 16 where scores of 0 to 6, 7 to 9 and 10 to 12 correspond to mild, moderate and severe spasticity respectively.
Post test Reaching Performance Scale | Change from baseline after 3 week treatment intervention
  Reaching Performance Scale (RPSS; Levin et al., 2004) evaluated performance of reaching and grasping tasks to objects placed within (RPSSnear) and beyond (RPSSfar) arm's length. Performance of 6 movement components is scored on 4-point (0-3) scales, for a total of 18 points per task. The RPSS scores correlate significantly with those of the Chedoke-McMaster Stroke Assessment and the Upper Extremity Performance Test for the Elderly (TEMPA) and discriminate between patients with different upper limb impairment levels. In addition, it was found to have good interrater reliability (67%).
Post test Box and Blocks Test | Change from baseline after 3 week treatment intervention
  Box and Blocks Test (BBT; Mathiowetz et al., 1985) is a functional dexterity test that involves moving blocks from one side of a box to the other by passing them over a barrier. Performance is scored according to the number of blocks transferred in 1 minute with lower scores corresponding to greater upper limb impairments. The BBT has high test-retest (Interclass Correlation Coefficient =0.94 - 0.98; Cromwell, 1976; Canny et al., 2009) and interrater (Interclass Correlation Coefficient =1.00) reliability.
Post test Motor Activity Log | Change from baseline after 3 week treatment intervention
  Motor Activity Log (MAL; Uswatte et al., 2006) is a structured questionnaire designed to assess the self-perceived use of the more-impaired arm after stroke while performing a wide range of basic and instrumental activities of daily life. Each item is scored on a 6 point scale (0 - 5). The scale has high internal consistency (Chronbach's α=0.87-0.95) and discriminative validity and highly correlates with caregiver responses (Interclass Correlation Coefficient = 0.52, p<0.05) and accelerometer recordings of actual arm use (r=0.7, p<0.05; Uswatte et al., 2005; 2006).
upper limb kinematics | One week before start of intervention
  Rigid body segmental kinematics will be recorded from sets of 4 passive reflective markers (0.5 cm diameter spheres) attached to the trunk, upper arm and forearm segments. This will enable the computation of three translational and three rotational degrees of freedom per segment. Marker motion will be recorded with a calibrated 3 camera optoelectronic motion-capture system (ProReflex MCU-240, Qualisys) on suitable PC software (QMT, Qualisys, Göteborg, Sweden). Data collection (100 Hrtz, 2-5 second) will be triggered by movement of the hand.
Follow-up Fugl-Meyer Arm Scale | Change from baseline 4 weeks after end of treatment intervention
  Fugl-Meyer Arm Scale (FMA; Fugl-Meyer, 1975) was developed to assess active motor function after stroke, based on the stages of recovery described by Twitchell and Brunnstrom (Sanford et al., 1993). Movements are scored between 0-2 points, and the summary score ranges from 0 (complete paralysis) to 66 (full ROM). The assessment has high validity (Berglund and Fugl-Meyer 1986) and reliability (Duncan et al. 1983) composite test-retest = 0.98-0.99; Interclass Correlation Coefficient for interrater reliability=0.96, p<0.0001; internal reliability = 90.7%) (Wolf et al., 2001).
Follow-up Composite Spasticity Index | Change from baseline 4 weeks after end of treatment intervention
  Composite Spasticity Index (CSI, Levin and Hui-Chan, 1992) assessed phasic (tendon jerk, clonus) and tonic (resistance to stretch) reflex responses in the elbow flexors when the limb was stretched at a moderate speed (>100/second). The valid (Nadeau et al. 1997) and reliable (Goulet et al. 1996) composite score ranges from 0 to 16 where scores of 0 to 6, 7 to 9 and 10 to 12 correspond to mild, moderate and severe spasticity respectively.
Follow-up Reaching Performance Scale | Change from baseline 4 weeks after end of treatment intervention
  Reaching Performance Scale (RPSS; Levin et al., 2004) evaluated performance of reaching and grasping tasks to objects placed within (RPSSnear) and beyond (RPSSfar) arm's length. Performance of 6 movement components is scored on 4-point (0-3) scales, for a total of 18 points per task. The RPSS scores correlate significantly with those of the Chedoke-McMaster Stroke Assessment and the Upper Extremity Performance Test for the Elderly (TEMPA) and discriminate between patients with different upper limb impairment levels. In addition, it was found to have good interrater reliability (67%).
Follow-up Box and Blocks Test | Change from baseline 4 weeks after end of treatment intervention
  Box and Blocks Test (BBT; Mathiowetz et al., 1985) is a functional dexterity test that involves moving blocks from one side of a box to the other by passing them over a barrier. Performance is scored according to the number of blocks transferred in 1 min with lower scores corresponding to greater upper limb impairments. The BBT has high test-retest (Interclass Correlation Coefficient =0.94 - 0.98; Cromwell, 1976; Canny et al., 2009) and interrater (Interclass Correlation Coefficient =1.00) reliability.
Follow-up Motor Activity Log | Change from baseline 4 weeks after end of treatment intervention
  Motor Activity Log (MAL; Uswatte et al., 2006) is a structured questionnaire designed to assess the self-perceived use of the more-impaired arm after stroke while performing a wide range of basic and instrumental activities of daily life. Each item is scored on a 6 point scale (0 - 5). The scale has high internal consistency (Chronbach's α=0.87-0.95) and discriminative validity and highly correlates with caregiver responses (Interclass Correlation Coefficient = 0.52, p<0.05) and accelerometer recordings of actual arm use (r=0.7, p<0.05; Uswatte et al., 2005; 2006).

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel